CLINICAL TRIAL: NCT04677114
Title: Integrated Outpatient Treatment of Opioid Use Disorder and Severe Injection Related Infections
Acronym: BOPAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laura Fanucchi (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Laura Fanucchi, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 60903; 1R01DA048892 (NIH)
Record Dates: First submitted 2020-12-13; First posted 2020-12-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Drug Use; Opioid-use Disorder
Keywords: buprenorphine; outpatient; parenteral; antibiotic; OPAT; injection; infectious endocarditis; injection-related; infection
MeSH Terms: conditions — Opioid-Related Disorders; Endocarditis, Subacute Bacterial; Infections | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination; Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Outpatient Parenteral Antibiotic Therapy (OPAT) (Experimental): Patients with opioid use disorder (OUD) and severe, injection-related infections (SIRI) will be treated with buprenorphine and be discharged with outpatient parenteral antibiotic therapy (OPAT).
  Interventions: Drug: Buprenorphine and Outpatient Parenteral Antibiotic Therapy
- Treatment as Usual (TAU) (Active Comparator): Patients with OUD and severe, injection-related infections (SIRI) will receive usual care.
  Interventions: Drug: Buprenorphine and standard of care antibiotic treatment

INTERVENTIONS:
Drug: Buprenorphine and Outpatient Parenteral Antibiotic Therapy — Participants will be complete IV antibiotics with OPAT. All participants will receive buprenorphine treatment of OUD.
  Other Names: Suboxone or Sublocade
  Arms: Outpatient Parenteral Antibiotic Therapy (OPAT)
Drug: Buprenorphine and standard of care antibiotic treatment — All participants will receive treatment of OUD and the infection per usual clinical care.
  Other Names: Suboxone or Sublocade
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study will assess the efficacy of an integrated outpatient treatment model for persons with opioid use disorder and injection related infections. The investigators hypothesize that outpatient antibiotic treatment coupled with comprehensive treatment for opioid use disorder will demonstrate a safe and effective way to manage patients. Results could improve the current protocols for the treatment of individuals with opioid use disorder and severe infections.

ELIGIBILITY:
Inclusion Criteria:

* have opioid use disorder
* have a severe injection related infection requiring antibiotics
* willing to accept buprenorphine treatment
* anticipated to be discharged home
* require IV antibiotic therapy

Exclusion Criteria:

* stroke or cerebral mycotic aneurysms preventing aortic or mitral valve surgery
* fungal valve IE
* requiring in-patient rehabilitation
* current pregnancy
* hypersensitivity or allergy to buprenorphine
* class III or IV heart failure
* end-stage liver or renal disease
* any condition that may prevent the volunteer from safely participating in the study
* self-report of desire to inject into the PICC line
* pending legal action that could interfere with study participation
* unsafe or unstable environment precluding safe administration of IV antibiotics
* living more than a 60 minute drive outside of Lexington, KY

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Illicit Opioid Use | 12 weeks after hospital discharge
  Proportion of urine samples with negative urine drug screen for illicit opioid use

SECONDARY OUTCOMES:
Completion of Recommended IV Antibiotic Therapy | up to 12 weeks (duration of IV antibiotic course as determined by treating physician)
  Proportion of patients who completed of recommended IV antibiotic therapy
Abstinence From Illicit Opioid | 12 weeks after hospital discharge
  Self-reported number of days of illicit opioid abstinence
Abstinence from Injection Drug Use | 12 weeks after hospital discharge
  Self-reported number of days without injection use of any drug
Outpatient Treatment Retention | 12 weeks after hospital discharge
  Number of days patients remain in treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanucchi LC, Murphy SM, Surratt H, Kapadia SN, Walsh SL, Grubbs JA, Thornton AC, Nuzzo P, Lofwall MR. Design and protocol of the Buprenorphine plus Outpatient Parenteral Antimicrobial Therapy (B-OPAT) study: a randomized clinical trial of integrated outpatient treatment of opioid use disorder and severe, injection-related infections. Ther Adv Infect Dis. 2022 Jul 11;9:20499361221108005. doi: 10.1177/20499361221108005. eCollection 2022 Jan-Dec. PMID 35847566

DOCUMENTS (1):
  • Informed Consent Form (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT04677114/ICF_000.pdf